CLINICAL TRIAL: NCT02544347
Title: Effects of Non-Surgical Periodontal Treatment on the Gingival Crevicular Fluid Levels of Vaspin and Omentin-1 in Type 2 Diabetic Patients With Chronic Periodontitis
Brief Title: Gingival Crevicular Fluid Vaspin and Omentin Levels in Type 2 Diabetic Patients With Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Asisstant Proffessor, Bulent Ecevit University, Bulent Ecevit University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-116-17/06
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Periodontitis; Diabetes Mellitus
Keywords: vaspin; omentin; diabetes mellitus; chronic periodontitis; tumor-necrosis factor alfa; gingival crevicular fluid
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- diabetes mellitus group (Other): gingival crevicular fluid was collected
  Interventions: Other: gingival crevicular fluid
- Control group (Other): gingival crevicular fluid was collected
  Interventions: Other: gingival crevicular fluid
- diabetics with chronic periodontitis group (Other): non-surgical periodontal treatment was completed and gingival crevicular fluid was collected
  Interventions: Other: gingival crevicular fluid; Other: non-surgical periodontal treatment
- chronic periodontitis group (Other): non-surgical periodontal treatment was completed and gingival crevicular fluid was collected
  Interventions: Other: gingival crevicular fluid; Other: non-surgical periodontal treatment

INTERVENTIONS:
Other: gingival crevicular fluid — gingival crevicular fluid was collected
Other: non-surgical periodontal treatment — scaling and root planing were performed
  Arms: chronic periodontitis group; diabetics with chronic periodontitis group

SUMMARY:
The aim of the present study were 1) to determine the role of these adipokines in the pathogenesis of periodontal disease, inflammation and tissue destruction comparing with gingival crevicular fluid (GCF) levels of TNF-α, which has a known pro-inflammatory effect in periodontal disease, 2) to investigate the effect of non-surgical periodontal treatment on GCF vaspin and omentin levels in type 2 diabetic (T2DM) patients with Chronic Periodontitis (CP).

DETAILED DESCRIPTION:
Adipose tissue produces and releases a variety of inflammatory factors, including adipocytokines , such as adiponectin, leptin, tumor-necrosis factor alpha (TNF-α), interleukin-6 (IL-6), visfatin, vaspin and omentin.These adipokines have widespread effects on carbohydrate and lipid metabolism and appear to play an important role in the pathogenesis of insulin resistance, diabetes, inflammation, wound healing, and immune responses.Recently, studies evaluated the serum vaspin and omentin levels as inflammatory markers in T2DM patients. Based on the above mentioned studies, the present investigation has been devoted to elucidate the role of adipokines in the pathogenesis that might link DM and periodontal disease. We hypothesize that vaspin and omentin are inflammatory adipokines involved in chronic inflammation and are associated with T2DM and CP. Additionally, the evaluation of GCF vaspin and omentin levels can provide advance the biologic link between DM and periodontitis. Until now, levels of GCF vaspin and omentin in CP patients with T2DM before and after non-surgical periodontal treatment has not been explored. Hence, the aim of the present study were 1) to determine the role of these adipokines in the pathogenesis of periodontal disease, inflammation and tissue destruction comparing with GCF levels of TNF-α, which has a known pro-inflammatory effect in periodontal disease 2) to investigate the effect of non-surgical periodontal treatment on GCF vaspin and omentin levels in T2DM patients with CP.

A total of 15 T2DM patients with CP ( DM-CP group), 15 CP patients (CP group), 15 T2DM patients (DM-CTRL group) and 15 subjects with systemically and periodontally healthy control subjects (CTRL group) were included in the study. Diabetic subjects should have T2DM and had no any known systemic diseases other than T2DM. The glycemic status of patients previously diagnosed with T2DM was confirmed by their glycated haemoglobin (HbA1c) levels. Periodontal disease status was determined according to clinical and radiographic criteria by the 1999 classification of periodontal disease.

Subjects were clinically evaluated using the following parameters; plaque index (PI), gingival index (GI) , PD, clinical attachment level (CAL) and BOP (deemed positive if it occurred within 15 seconds after probing). Clinical measurements were recorded by one calibrated examiner at six sites per tooth from the full-mouth teeth excluding third molars using with a Williams periodontal probe (Nordent Manufacturing Inc., ElkGrove Village, IL, USA) calibrated in millimeters. Anthropometric measurements included weight (kg) and height (m) of the subjects to calculate the BMI ( weight divided by the square of height, kg/m2 ).

All clinical and radiological examinations, sampling site selections were performed by one examiner and the samples were collected on the day after clinical examination of patients. This was to prevent contamination of GCF with blood associated with the probing of inflamed sites. The deepest two pocket sites of single-rooted teeth were selected for the collection of GCF in both periodontitis groups, and also two pocket sites with an absence of inflammation were sampled to ensure the collection of an adequate amount of GCF in control groups. In patients from CP and DM-CP groups, sites showing greatest PD when measured with a periodontal probes and signs of inflammation, along with radiographic conformation of bone loss were sampled. GCF samples were collected at baseline and after 8 weeks from baseline sampling in both periodontitis groups, and only at baseline in control groups. To avoid salivary contamination, the sites to be sampled were rinsed with water, isolated by cotton rolls and gently air dried. Paper strips (Periopaper; Oraflow Inc.,Smithtown, NY, USA) were gently inserted 1-2 mm into the sulcus/pocket for 30 seconds. Care was taken to avoid mechanical injury of the gingival tissues. All samples containing blood and saliva were discarded. The two strips from two sites of each individual were placed into coded sealed plastic eppendorf tubes and pooled before freezing at -80 degree

ELIGIBILITY:
Inclusion Criteria:

* Diabetic subjects should have T2DM and had no any known systemic diseases other than T2DM
* Subjects who had HbA1c levels < 8% and ≥ 6.5% (well and moderate control)
* Chronic periodontitis patients had radiographic evidence of bone loss and attachment loss with a minimum of 6 teeth having pocket probing depth (PD) ≥ 5mm in at least 2 different quadrants
* Control groups were designed as healthy if the full-mouth probing depth (PD) was ≤3mm and bleeding on probing (BOP) score < %15 at examination and they had no radiographic evidence of alveolar bone loss.

Exclusion Criteria:

* Presence of other systemic disorders that could influence the course of periodontal disease; pregnancy, lactation, current and former use of tobacco;
* Administration of non-steroidal and anti-inflammatory drugs or antibiotic therapies within the previous 6 months;
* Need for antibiotic prophylaxis for dental treatment and having received non-surgical periodontal treatment within the past 6 months or surgical periodontal treatment within the past 12 months.
* Subjects who had body mass index (BMI) >24.9 kg /m2

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
vaspin levels | 8th weeks
  gingival crevicular fluid vaspin levels change from baseline at 8th weeks
omentin levels | 8th weeks
  gingival crevicular fluid omentin levels change from baseline at 8th weeks

SECONDARY OUTCOMES:
tumor necrosis factor alfa | 8th weeks
  change of gingival crevicular fluid tumor necrosis factor alfa levels from baseline at 8th weeks
gingival index | 8ths week
  gingiva inflammation score
plaque index | 8th weeks
  oral hygen score
bleeding on probing | 8th weeks
  deemed positive if it occurred within 15 seconds after probing
clinical attachment level | 8th weeks
  distance between the cemento-enamel junction to the deepest point of periodontal pocket

CONTACTS AND LOCATIONS:
Overall Officials: Umut Ballı, DDS, Principal Investigator — Bülent Ecevit University Faculty of Dentistry; Şeyma Bozkurt Doğan, DDS, Study Chair — Bülent Ecevit University Faculty of Dentistry; Figen Öngöz Dede, DDS, Principal Investigator — Bülent Ecevit University Faculty of Dentistry; Erdim Sertoğlu, MD, DDS, Principal Investigator — Gülhane Military Medical Academy